CLINICAL TRIAL: NCT03888521
Title: Evaluating the GN ReSound Relief App Using task-and Rest-based fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: GN Hearing A/S (Industry)
Responsible Party: Principal Investigator, Fatima Husain, Associate Professor, Department of Speech and Hearing Science, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18895
Record Dates: First submitted 2019-03-18; First posted 2019-03-25 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Tinnitus, Subjective
Keywords: Relief
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Efficacy of a non-invasive intervention is being tested, while exploratory data is also being collected to better understand tinnitus
Masking Description: All participants receive the intervention, serving as their own controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resound Relief (Experimental): All participants are in the same group, and receive the same intervention - use of the Resound Relief smartphone app for 6 months
  Interventions: Behavioral: Resound Relief smartphone app

INTERVENTIONS:
Behavioral: Resound Relief smartphone app — The intervention is a smartphone app which has been developed to include a wide range of sounds and techniques aimed at reducing the impact of tinnitus.

SUMMARY:
The main goal of this study is to assess the effectiveness of the Resound Relief app in alleviating problems associated with tinnitus, using both behavioral assessment and brain imaging. Subjective tinnitus ("ringing in the ears") is the false perception of sound in the absence of an external stimulus. It often causes emotional distress and, in severe cases, interferes with daily activities and can lead to anxiety and depression. Sound therapy and relaxation techniques have been widely used as prominent interventions to ameliorate the adverse effects of tinnitus on overall health and psychological variables. The Resound Relief app combines the merit of these two kinds of therapy to allow the patients to alternate between therapies and manipulate them according to their specifics and needs. To assess the efficacy of the Resound Relief app in relieving tinnitus, the investigators will perform an interventional study in which tinnitus patients will use the app installed on their smart phones for six months. The effects of this intervention will be quantified via audiological and cognitive assessments, administering questionnaires and surveys, and MRI scanning sessions. Audiological and cognitive assessments, and MRI scanning will be conducted before and six months after the use of the Resound Relief app. Tinnitus-related questionnaires will be administered before, two, four, and six months after beginning use of the app. A short survey will be filled out every week regarding participants' experience with the app, tracking changes in the users' tinnitus, hearing loss and general emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* Screening questionnaires:

  * Tinnitus and Hearing Healthcare History (THH) form: This form is intended to assess subjects' healthcare history. The manner in which it is used to exclude subjects due to health issues other than tinnitus and hearing loss is described in the exclusion criteria.

For the purpose of this study (i.e. intervention), the investigators will include participants with managed depression or anxiety, as it may be difficult to recruit participants with severe tinnitus that do not have one or both of those conditions. However, only subjects aged between 21- 70 years old will be included.

* Tinnitus Functional Index (TFI): The investigators will recruit participants with varying degrees of tinnitus severity, reflecting the real-world usage of the app, but with a preference that at least 50% of the subjects have bothersome tinnitus defined as greater than 25 on the TFI scale (0-100).
* Audiometric evaluation (described in research procedures): The audiometric evaluation will primarily be used to obtain participants' hearing profiles. Subjects who have normal hearing thresholds (defined as less than or equal to 30 dB HL) up to 1 kHz in at least one ear will be included. Subjects who do not meet the defined normal hearing thresholds will be assessed on a case by case basis to ensure they can communicate without assistance with the investigators during scanning.

Exclusion Criteria:

* Screening questionnaires:

  * Tinnitus and Hearing Healthcare History (THH) form: This form contains questions regarding confounding variables such as traumatic brain injury (TBI), post-traumatic stress disorder, Ménière's disease, drug and alcohol use, and neurological or psychiatric health issues such as epilepsy. In the event that a participant has any of the described conditions or uses drugs/drinks to excess, those participants will be excluded from the study.

Drug/alcohol abuse will be assessed by questions 31 and 32 in the THH Form. If a subject indicates 'yes' to question 32, indicating that they have abused drugs or alcohol within the last 2 years, those participants will be excluded from the study. Studies have shown that a history of drug or alcohol abuse affects brain patterns as measured by MRI. Because the investigators need to average in order to report our results, outliers can change our results. For this reason, the investigators ask question 31 regarding past drug and alcohol use to better understand our data set. Exclusion, however, will only be based on usage within the last 2 years (question 32). The questionnaire also asks for a list of medications currently being used; some are known to affect tinnitus, and participants using such medications will be excluded.

* BDI and BAI: If a subject presents with significant depression and/or anxiety those participants will be excluded. This is demonstrated via a score above 30 on the Beck Depression Inventory (BDI) and/or above 25 on the Beck Anxiety Inventory (BAI). Further, the BDI contains a question (#9) asking about suicidal thoughts. This question will not be asked and has been deleted from the questionnaire given to the subjects.
* Mini-Mental State Examination: Participants will be excluded from the study if they do not have normal cognition, i.e. if a given score of 27 out of 30 or lower is achieved on the Mini-Mental State Examination.
* BIC safety screening form: This questionnaire contains questions regarding claustrophobia and whether there are any metal implants or pieces (such as metal flakes in the eyes from metal work) that may pose a health risk under the strong magnetic fields used in MRIs. Participants that indicate having metal in their bodies will be excluded. Those that indicate claustrophobia will be assessed for inclusion via the mock scan (see below).

  * Audiometric evaluation:
* Participants with hearing aids will be evaluated on a case-by-case basis as to their communication abilities without hearing aids.
* Loudness Discomfort Level: Loudness Discomfort Levels (LDLs) measured during the assessment will be used to verify whether participants will be able to tolerate the noise level of the scanner. Hearing protection will be provided during the MRI scans; however, participants with low LDLs may still experience discomfort. For their comfort, if participants report that a sound is uncomfortable at an LDL of 75 dB HL or quieter, those participants will be excluded from the MRI scanning portion of the study. If a participant has an LDL between 76 and 90 dB HL, they will be assessed on a case by case basis for comfort within the MRI scanner (the investigators will play scanner noise for the participants, take into consideration any past MRIs participants have had, etc.). If participants have an LDL of 90 dB HL or higher, those participants will be able to tolerate the noise level of the scanner and will be included.

  * MRI Scans (described in research procedures):
* Mock scan: If participants meet the above criteria, they will be asked to complete a mock MRI scan. During this mock scan, participants will be placed inside a non- operational model of the MRI magnet to verify they are not claustrophobic and will be comfortable during the MRI scans.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduced tinnitus annoyance measured via Tinnitus Functional Index | baseline, 2 months, 4 months and 6 months
  The Tinnitus Functional Index (TFI) is a tinnitus questionnaire, widely used to quantify tinnitus annoyance. It contains 25 questions, each of which participants rate from a scale of 0-10. The scores are then averaged, to give an overall score from 0 to 100. Higher values indicate higher disturbance and annoyance from tinnitus.
  There are also 8 subscales in the questionnaire, which are each also averaged to give scores from 0 to 100. The subscales look at various aspects of tinnitus annoyance, specifically (1) intrusiveness, (2) reduced sense of control, (3) cognitive interference, (4) sleep disturbance, (5) auditory difficulties, (6) interference with relaxation, (7) reduced quality of life and (8) emotional distress.
  The questionnaire will be completed by participants before (baseline), and 2, 4 and 6 months after using the app for a minimum of 1 hour a day, 5 days a week. The investigators hope to see reduction in the reported annoyance of tinnitus in participants' lives.
Reduced tinnitus annoyance measured via Iowa Tinnitus Primary Function Questionnaire | baseline, 2 months, 4 months and 6 months
  The Tinnitus Primary Function Questionnaire (TPFQ) is a tinnitus questionnaire, widely used to quantify tinnitus annoyance. It contains 20 questions, each of which participants rate from a scale of 0-100. The scores are then averaged, to give an overall score from 0 to 100. Higher values indicate higher disturbance and annoyance from tinnitus.
  There are also 4 subscales in the questionnaire, which are each also averaged to give scores from 0 to 100. The subscales look at various aspects of tinnitus annoyance, specifically (1) difficulties in concentration, (2) emotional distress, (3) hearing difficulties, and (4) sleep difficulties.
  The questionnaire will be completed by participants before (baseline), and 2, 4 and 6 months after using the app for a minimum of 1 hour a day, 5 days a week. The investigators hope to see reduction in the reported annoyance of tinnitus in participants' lives.
Reduced tinnitus annoyance measured via Tinnitus Handicap Inventory | baseline, 2 months, 4 months and 6 months
  The Tinnitus Handicap Inventory (THI) is a tinnitus questionnaire, widely used to quantify tinnitus annoyance. It contains 25 questions, each of which participants rate one of "Yes," "Sometimes," or "No." Any "Yes" response is scored as 4 points, "Sometimes" is scored as 2 points, and "No" is scored as 0 points. The totals are then added up, giving an overall questionnaire score that can range from 0-100. Higher values indicate higher disturbance and annoyance from tinnitus.
  The questionnaire will be completed by participants before (baseline), and 2, 4 and 6 months after using the app for a minimum of 1 hour a day, 5 days a week. The investigators hope to see reduction in the reported annoyance of tinnitus in participants' lives.

SECONDARY OUTCOMES:
Analyzing changes in neural gray matter using voxel-based morphometry (VBM) | baseline, and 6 months
  Voxel-based morphometry (VBM) is a computational analytical technique that measures differences in local concentrations of brain tissue. VBM is applied to high-resolution anatomical images collected via magnetic resonance imaging. The unit of this measurement is mm3 of original grey matter per mm3 of spatially normalised space within the participant's brain image.
  Whole-brain VBM comparisons will be applied within each participant's data, comparing their total gray matter brain volume before use of the smartphone app to total gray matter brain volume after 6 months of using the app.
Analyzing changes in neural white matter using diffusion tensor imaging (DTI) | baseline, and 6 months
  Diffusion tensor imaging (DTI) is a magnetic resonance imaging technique which enables the measurement of the movement of water molecules within tissue, allowing us to track a white matter tract and calculate its microstructural integrity.
  Fractional anisotropy (FA), which is a scalar value ranging from 0 to 1, is a DTI measure which allows us to calculate how freely the water molecules within a measured tissue can move. Tractography is a modeling technique used to visually represent nerve tracts within the brain, which is derived from the DTI data collected.
  FA will be calculated, and tractography modeled, for each participant, comparing their total white matter microstructural integrity before use of the smartphone app and after 6 months of using the app.
Analyzing changes in resting state neural networks using functional magnetic resonance imaging | baseline, and 6 months
  Resting state functional connectivity is a functional magnetic resonance imaging technique used to evaluate interactions between various brain regions while the brain is at waking rest. The technique measures the haemodynamic response of the brain after magnetic pulses are sent by the scanner. This response is measured on a scale known as the Blood Oxygen Level Dependent (BOLD) signal, which is relative. Correlations of activity seen between brain regions is believed to be indicative of neural networks.
  The resting state functional connectivity will be measured for each participant, before, and after 6 months of using the app.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Husain, PhD, Principal Investigator — University of Illinois at Urbana-Champaign, Department of Speech and Hearing Science
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No